CLINICAL TRIAL: NCT06434246
Title: Effect of Pully System Exercise on Upper Limb Function in Hemiplegic Cerebral Palsy Children: a Randomized Clinical Trials
Brief Title: Effect of Pully System on Hemiplegic Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Ali Mohammed Torad, Lecturer, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200--194
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): 16 Children will undergo a pulley system exercise regimen tailored to improve upper limb function in addition to designed physical therapy program for CP.
  Interventions: Behavioral: pulley system exercise regimen; Biological: physical therapy program for CP
- Control Group (Active Comparator): Children will receive designed physical therapy program for CP only
  Interventions: Biological: physical therapy program for CP

INTERVENTIONS:
Behavioral: pulley system exercise regimen — The warm-up consists of gentle stretching and basic mobility exercises to prepare the muscles and joints for the activity. Following this, the main segment of the session involves specific exercises using the pulley system, designed to target and improve motor function, strength, and coordination of the upper limbs. The therapist will adjust the exercises according to each child's individual abilities and progression over time. The session concludes with a cool-down period involving light activities and relaxation techniques to ensure a gradual return to baseline physiological states.
  Arms: Intervention Group
Biological: physical therapy program for CP — Participants in the control group will attend physical therapy sessions twice per week. These sessions aim to maintain or improve physical functioning and manage the symptoms of cerebral palsy. Each session lasts approximately 45 to 60 minutes, These sessions include a variety of therapeutic exercises tailored to each child's needs but do not include the use of the pulley system. Typical activities might involve stretching, strengthening exercises, and manual therapy techniques to enhance joint mobility and muscle function.

SUMMARY:
Introduction Cerebral palsy (CP) is a group of sensory, motor, and postural disorders caused by non-progressive brain injury in early development. It can manifest in various forms, including hemiplegia, which affects about 21% to 40% of CP cases. Upper extremity (UE) impairments in CP individuals are significant, impacting daily activities and quality of life.

Objective This study aims to investigate the effects of pulley system exercises on improving upper limb function in children with hemiplegic CP.

Methods Design: Randomized controlled double-blinded trial. Participants: 32 children aged 3-7 years with hemiplegic CP, divided into intervention and control groups.

Intervention: The intervention group receives pulley system exercises plus standard care, while the control group receives standard physical therapy.

Duration: Conducted between June 2024 and August 2024. Inclusion Criteria: Diagnosed with hemiplegic CP, aged 3-7 years, able to follow instructions, and with upper limb motor deficits.

Exclusion Criteria: Additional neurological disorders, recent upper limb surgery, previous rehabilitation programs, severe medical conditions, or contraindications to physical activity.

Assessment Tools: Assisting Hand Assessment (AHA), Bruininks-Oseretsky Test of Motor Proficiency (BOT-2), Quality Upper Extremity Skills Test (QUEST), and Lafayette Manual Muscle Tester.

Timing: Baseline and after 3 months of intervention. Treatment Intervention Group: 45-60 minute sessions, three times a week, involving warm-up, pulley system exercises, and cool-down.

Control Group: Standard care physical therapy, twice a week, 45-60 minute sessions.

Statistical Analysis Methods: Descriptive statistics and Analysis of Covariance (ANCOVA) to analyze improvements in upper limb function.

Significance Level: p < 0.05. Analysis: Intention-to-treat to handle missing data. This study aims to provide evidence on the effectiveness of pulley system exercises in enhancing upper limb function in children with hemiplegic CP, potentially improving their independence and quality of life.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a collection of sensory and motor disorders, as well as postural disorders, caused by non-progressive injury to the immature brain1,2. It can be classified according to the topographical presentation as monoplegia, hemiplegia, diplegia, and quadriplegia2 . These obvious motor difficulties are frequently accompanied by cognitive disturbances and other neurologic difficulties3 . CP is considered the most prevalent mobility disorder in children, with an average frequency of 3 per 1,000 live births worldwide and a high prevalence of 60 to 150 per 1,000 among preterm infants who are born weighing less than 1,500 g 4 . Hemiplegic CP accounts for 21% to 40% of all cases of CP5,6.

Impairments in the upper extremity (UE) are a major factor for activity limitation and participation restriction in individuals with CP and may affect up to 50% of CP subjects [7]. UE limitations are mostly due to a lack of trunk control, decrease in shoulder girdle motor control and imbalance between spastic and paretic muscles [8]. That makes it difficult for people with CP to perform UE-specific tasks, such as reaching, grasping and manipulation, and it leads to the significant involvement of the positioning and functioning of the elbows, wrists and hands . Moreover, a lack of autonomy and dependence on other people may affect the individuals' quality of life [9].

Pulley therapy is a part of universal exercise unit which formed of spider cage and a system of pulley, straps and weights for resistance. It is a new method used for strengthening of weak muscles by isolating the target specific muscle for training [10] . There are several benefits of pulley therapy as: improving passive/active ROM, flexibility of muscle, enhancing strength and endurance of muscle without any associated movement and improving functional skills and dynamic movement [11] .

So, this study was conducted to investigate the effect of pully system exercise in improvement of upper limb function in hemiplegic cerebral palsy children

Subjects materials and methods:

Randomized controlled double blinded study design was used. The study will be conducted at El salam university out- patient clinic between June 2024 and August 2024 Subjects G power v2.1.9.7 was used to calculate proper sample size based on pilot testing that revealed effect size of 1.05. the proposed sample size is 32 when using alpha of 0.05 and power of 80%.

The sample size will equal 32 (randomly divided into two group) study group will receive poly system exercise on upper limb, Control group will receive designed physical therapy programme.

Once participants meet the inclusion criteria and consent to participate, they are randomly assigned to either the intervention group (receiving pulley system exercises in addition to standard care) or the control group (receiving standard care). Use a computer-generated random number table or software to assign participants.

The therapists or researchers who conduct the evaluations (e.g., AHA, BOT-2, QUEST) will not be informed of the participant's group assignment. This can be achieved by using different individuals to provide the intervention and assess the outcomes, or by ensuring that assessment data are coded in such a way that the assessor does not know the group codes.

Participants will be randomly assigned to one of two groups:

Group (A): Intervention Group: 16 Children will undergo a pulley system exercise regimen tailored to improve upper limb function in addition to designed physical therapy program for CP.

Group (B): Control Group: Children will receive designed physical therapy program for CP only.

ELIGIBILITY:
Inclusion Criteria

* Children aged between 3 and 7 years.
* Diagnosed with hemiplegic cerebral palsy, confirmed by a pediatric neurologist.
* Ability to follow simple instructions and participate in exercise sessions.
* Presence of upper limb motor function deficits attributable to hemiplegic cerebral palsy.

Exclusion Criteria

1. Children with additional neurological disorders or severe cognitive impairments that might interfere with the ability to participate in exercise regimens.
2. Recent surgery (within the last 6 months) on the upper limbs.
3. Children who have been involved in similar rehabilitation programs in the past 3 months.
4. Severe uncontrolled medical conditions such as cardiac or respiratory diseases. Presence of any contraindication to physical activity as advised by a medical professional.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Assisting Hand Assessment (AHA) | 3 months
  will be used to evaluate how effectively children with upper limb impairments can use their affected hand together with their well-functioning hand to perform bimanual tasks. This assessment involves observing the child while they engage in play activities that require bimanual coordination. The performance is video-recorded and scored based on specific criteria that assess the spontaneous use of the involved hand. The scoring system provides a measure of the child's ability to effectively use their affected hand in bimanual tasks, with higher scores indicating better function.
The Bruininks-Oseretsky Test of Motor Proficiency (BOT-2) for Hand Function | 3 months
  will be conducted to measures fine and gross motor skills, including hand function. Specific subtests related to hand function are administered, such as fine motor precision, fine motor integration, and manual dexterity tasks. Performance on these tasks is quantitatively scored, allowing for the assessment of motor proficiency and hand function improvements
Quality Upper Extremity Skills Test (QUEST) | 3 months
  will be used to assess movement patterns and hand function in children with cerebral palsy. It evaluates dissociated movements, grasp patterns, protective extension, and weight bearing under four domains: dissociated movements, grasp, weight bearing, and protective extension. Each item is scored based on the child's ability to perform the task, with scores reflecting the quality of upper extremity skills.
Lafayette Manual Muscle Tester | 3 months
  will be used to objectively measure the strength of specific muscles and muscle groups. The muscle tester is applied to the muscle group being evaluated while the child performs a muscle contraction. The device provides a digital readout of the force exerted, which can be measured in pounds or kilograms. In this study, the tester will be used to evaluate the strength of upper limb muscles before and after the intervention to assess any changes due to the pulley system exercises

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed salim, PHD, Study Director — Department of pediatric physical therapy and its surgery, Elsalam University; Sara Elsebahy, PHD, Study Director — Paediatric physical therapy department, Kafrelsheik University; Ahmed Ali M Torad, PHD, Principal Investigator — Basic science department, kafrelsheik university
Locations (1):
- Faculty of physical therapy, Kafrelsheik university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data to be Shared: The de-identified individual participant data that will be shared includes baseline demographic information, outcome measures from the Assisting Hand Assessment (AHA), Bruininks-Oseretsky Test of Motor Proficiency (BOT-2), Quality Upper Extremity Skills Test (QUEST), and muscle strength data from the Lafayette Manual Muscle Tester. This also includes data on the intervention details such as session frequency, duration, and adherence.
  Time Frame: Data will be available for sharing beginning 6 months after the publication of the study results. The data will be accessible for a period of 5 years.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing beginning 6 months after the publication of the study results. The data will be accessible for a period of 5 years.
Access Criteria: Researchers who wish to access the data must submit a formal request to the principal investigator. The request should include a research proposal outlining the purpose of the data use, the intended analysis, and the potential benefits of the research. Requests will be reviewed based on scientific merit and ethical considerations.